CLINICAL TRIAL: NCT03276286
Title: A Feasibility Study of the Nativis Voyager® System in Patients With Newly Diagnosed Glioblastoma Multiforme (GBM)
Brief Title: Nativis Voyager for Newly Diagnosed GBM
Acronym: NAT109
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nativis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NAT109
Record Dates: First submitted 2017-09-05; First posted 2017-09-08 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Nativis Voyager combined with standard radiotherapy and temozolomide
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Nativis Voyager (Experimental): Nativis Voyager combined with SOC Radiotherapy and temozolomide
  Interventions: Device: Nativis Voyager

INTERVENTIONS:
Device: Nativis Voyager — Nativis Voyager treatment combined with standard of care radiotherapy and temozolomide

SUMMARY:
This feasibility study will assess the effects of the Nativis Voyager therapy in patients newly diagnosed with GBM. The study will enroll and treat up to 32 subjects and will be combined with standard of care radiotherapy and temozolomide.

ELIGIBILITY:
Inclusion Criteria:

* There is pathological evidence of GBM using World Health Organization (WHO) classification.
* Subject received maximal debulking surgery. Patients may enroll in the study if received Gliadel wafers before entering the trial. Any additional treatments received prior to enrollment will be considered an exclusion.
* Subject must have at least one measurable lesion per RANO.
* Subject is at least 18 years of age.
* Subject has a Karnofsky Performance Scale (KPS) ≥ 60.
* Subject has life expectancy > 3 months.
* Subject has adequate organ and marrow function; see note 1.
* Subject able to start treatment at least 28 days from tumor resection surgery.
* Subject has provided signed informed consent.

Exclusion Criteria:

* Subject has progressive disease per RANO. If pseudoprogression is suspected, additional imaging studies must be performed to rule out true progression.
* Evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness)
* Subject is currently being treated with Optune.
* Subject is currently being treated with other investigational agents.
* Subject has not sufficiently recovered from prior surgery in the opinion of the investigator.
* Subject has significant co-morbidities at baseline which would prevent radiotherapy and/or temozolomide treatment.
* Subject has history of hypersensitivity reaction to temozolomide or a history of hypersensitivity to dacarbazine (DTIC).
* Subject has a clinically significant electrolyte abnormality.
* Subject has an active implantable (e.g., neurostimulator, pacemaker) or other electromagnetic device that is incompatible with MRI. Subjects with programmable shunt are excluded from the study.
* Subject has a metal implant, including a stent, in the head or neck that is incompatible with MRI.
* Subject is known to be HIV positive.
* Subject is pregnant, nursing or intends to become pregnant during the study period.
* Subject is participating in other potentially confounding investigational research.
* Subject has any condition that at the discretion of the investigator would preclude participation in the study.
* Subject is unable or unwilling to comply with the protocol-required follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Treatment-related Adverse Events (Safety) | Through study completion, average of 1 year
  Safety as measured by number of investigational treatment-related adverse events as assessed by CTCAE v4.0.

SECONDARY OUTCOMES:
Clinical Utility PFS | 6 months
  Progression Free Survival
Clinical Utility OS | Through patient completion, expected average 8 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Donna Morgan Murray, PhD, Study Chair — Nativis, Inc.
Locations (7):
- United States (7):
  - Center for Neurosciences, Tucson, Arizona
  - California Cancer Care Associates, Encinitas, California
  - John Wayne Cancer Institute @ Providence St Johns Health Center, Santa Monica, California
  - Associated Neurologists of Southern CT, PC, Fairfield, Connecticut
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Cancer Care Collaborative, Austin, Texas
  - Baylor Scott and White Health, Temple, Texas

IPD SHARING:
Plan to Share IPD: No